CLINICAL TRIAL: NCT04941482
Title: Intervention Effectiveness Towards Improving Physical and Mental Health for Post-stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: National Geriatric Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 9720701; 494/GCN-HDDDNCYSH-DHYHN (Other: Hanoi Medical University Institutional Ethical Review Board)
Record Dates: First submitted 2021-06-10; First posted 2021-06-28 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Brain Infarction; Brain Ischemia; Cerebral Infarction; Cerebrovascular Disorders
Keywords: Stroke; Mental Health; Physical activity; Cognitive therapy; Motivational Interviewing; fNIRs; Functional near-infrared spectroscopy; Rehabilitation
MeSH Terms: conditions — Stroke; Brain Infarction; Brain Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Psychological Well-Being; Motor Activity | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: 92 stroke patients registered at the Vietnam National Geriatrics Hospital were enrolled in the study for 6 months. The patients were randomly assigned to either an intervention group that received the long-term follow-up program, or a control group that received standard care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-intervention program (Experimental): A multi-intervention program was designed for stroke patients, including: [1] periodic health examinations for assessing physical and mental health, recurrence risks, and harmful behaviors; [2] guiding appropriate rehabilitation exercises to improve physical status and monitoring through daily online reports; [3] using motivational interviewing methods to improve and prevent mental disorders; [4] using the technique of functional near-infrared spectroscopy (fNIRS) to measure oxy-hemoglobin in the prefrontal cortex to early detect mental disorders and stroke recurrence risks.
  Interventions: Behavioral: Periodic health check program for post-stroke; Behavioral: Guiding the appropriate rehabilitation exercises; Behavioral: Motivational Interviewing; Device: Functional near-infrared spectroscopy
- Standard care (Active Comparator): The control group received the standard health check and was measured by an fNIRS device.
  Interventions: Behavioral: Periodic health check program for post-stroke; Device: Functional near-infrared spectroscopy

INTERVENTIONS:
Behavioral: Periodic health check program for post-stroke — The stroke survivors were assessed for their physical and mental health, recurrence risks, and harmful behaviors at 0, 1, 3, and 6 months using specific scales.
Behavioral: Guiding the appropriate rehabilitation exercises — The appropriate rehabilitation exercises were designed and guided for each patient, and they were followed up by the daily online report.
  Arms: Multi-intervention program
Behavioral: Motivational Interviewing — Motivational Interviewing will carry out on post-stroke patients in the first three months (one time per week in the first month and one time per the second and third month). This intervention method aims to discover and resolve patient's conflicts by a standardized communication skill to improve their mental health and change negative behaviors.
  Other Names: Cognitive therapy
  Arms: Multi-intervention program
Device: Functional near-infrared spectroscopy — The fNIRS devices served as an effective monitoring and therapeutic tool, evaluating the evolution of neural activity and stroke rehabilitation and recovery. Moreover, the cortex hemodynamic measurement by fNIRS could detect various mental disorders such as depression, anxiety, schizophrenia early through cognitive tasks.
  Other Names: fNIRS

SUMMARY:
This was a multi-intervention randomized controlled trial that aimed to develop a management pattern for stroke survivors. The program consisted of monitoring the recovery process, early detecting the physical and mental disorders, suitably intervening for each patient to improve their quality of life. New intervention techniques were firstly applied for post-stroke patients in Vietnam such as using the portable functional near-infrared spectroscopy (fNIRS) device to explore cortex frontal hemodynamic and motivational interviewing for psychological adjustment. A total of 92 stroke patients registered in Vietnam National Geriatrics Hospital were included in the study for 6 months. Included patients were randomized to an intervention group and received the long-term follow-up program or to a control group receiving standard care. The mental health and physical functioning of participants were assessed at 0, 1, 3, and 6 months follow-up. This work was funded by Vingroup Joint Stock Company and supported by the Domestic Master/Ph.D. Scholarship Programme of Vingroup Innovation Foundation (VINIF), Vingroup Big Data Institute (VINBIGDATA).

DETAILED DESCRIPTION:
Stroke is a medical condition that occurs when a blood vessel that carries oxygen and nutrients to the brain is either blocked by a clot or bursts (or ruptures). This is a major cause of death and disability worldwide. Post-stroke patients will experience sudden and intense changes in their physical and mental health during the first year. Currently, there is no official management model for improving the physical and mental health of patients after stroke in Vietnam. Furthermore, traditional neuroimaging techniques such as Functional magnetic resonance imaging (fMRI), Positron emission tomography (PET), Electroencephalogram (EEG) are not suitable for routine monitoring due to limited flexibility dynamics and costs. Hence, this study aimed to develop a management pattern that included monitoring the recovery process, early detecting the physical and mental disorders, suitably intervening for each patient to improve their quality of life. New intervention techniques were firstly applied for post-stroke patients in Vietnam such as using the portable fNIRS device to explore cortex frontal hemodynamic and motivational interviewing for psychological adjustment. This randomized controlled trial study included 92 post-stroke patients with dividing into two groups (46 control & 46 intervention subjects), who experienced emergency by stroke within one week. A multi-intervention program was designed for stroke patients including [1] periodic health examination for assessment of physical and mental health, recurrence risks, and harmful behaviors; [2] guiding the appropriate rehabilitation exercises for improving the physical status and monitoring through daily online reports; [3] using motivational interviewing methods to improve and prevent mental disorder; [4] application of the technique of functional near-infrared spectroscopy (fNIRS) for measurement of oxy-hemoglobin on cortex prefrontal to early detect mental disorder and stroke recurrence risks. Outcome data were collected via study questionnaires and fNIRS measuring results which were administered by researchers in the study site at 0, 1, 3, and 6 months follow-up. Simultaneously, Motivational Interviewing was carried out on post-stroke patients in the first three months (one time per week in the first month and one time per second and third month). This intervention method aimed to discover and resolve patient's conflicts by standardized communication skill to improve their mental health and change negative behaviors. The scores of the Stroke Impact Scale (SIS), physical and mental assessment scales and fNIRS data in both groups were used to calculate the effect estimates of intervention methods with a measure of precision (95% CI) and assess the results of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke according to WHO's definition of stroke
* Are managed at the National Geriatrics Hospital in Vietnam
* Include 24 hours to 1 week after stroke
* Provide informed consent
* Willing to attend intervention therapies & follow-up evaluations for half-year.
* Have conscious, cognitive, and communication abilities.

Exclusion Criteria:

* Do not agree to participate in the study
* Are included in other experimental studies
* Have mental disorders before stroke attack
* Glasgow score ≤ 8
* Other diseases that make it difficult to complete the intervention

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thao TP Nguyen, MD, MSc, Principal Investigator — Hanoi Medical University, Hanoi 100000, Viet Nam
Locations (1):
- National Geriatrics Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feigin VL, Roth GA, Naghavi M, Parmar P, Krishnamurthi R, Chugh S, Mensah GA, Norrving B, Shiue I, Ng M, Estep K, Cercy K, Murray CJL, Forouzanfar MH; Global Burden of Diseases, Injuries and Risk Factors Study 2013 and Stroke Experts Writing Group. Global burden of stroke and risk factors in 188 countries, during 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet Neurol. 2016 Aug;15(9):913-924. doi: 10.1016/S1474-4422(16)30073-4. Epub 2016 Jun 9. PMID 27291521
- [Background] Cheng D, Qu Z, Huang J, Xiao Y, Luo H, Wang J. Motivational interviewing for improving recovery after stroke. Cochrane Database Syst Rev. 2015 Jun 3;2015(6):CD011398. doi: 10.1002/14651858.CD011398.pub2. PMID 26037617
- [Background] Petersen TH, Willerslev-Olsen M, Conway BA, Nielsen JB. The motor cortex drives the muscles during walking in human subjects. J Physiol. 2012 May 15;590(10):2443-52. doi: 10.1113/jphysiol.2012.227397. Epub 2012 Mar 5. PMID 22393252
- [Background] Miyai I, Yagura H, Hatakenaka M, Oda I, Konishi I, Kubota K. Longitudinal optical imaging study for locomotor recovery after stroke. Stroke. 2003 Dec;34(12):2866-70. doi: 10.1161/01.STR.0000100166.81077.8A. Epub 2003 Nov 13. PMID 14615624
- [Background] Strangman G, Goldstein R, Rauch SL, Stein J. Near-infrared spectroscopy and imaging for investigating stroke rehabilitation: test-retest reliability and review of the literature. Arch Phys Med Rehabil. 2006 Dec;87(12 Suppl 2):S12-9. doi: 10.1016/j.apmr.2006.07.269. PMID 17140875
- [Background] Mihara M, Miyai I. Review of functional near-infrared spectroscopy in neurorehabilitation. Neurophotonics. 2016 Jul;3(3):031414. doi: 10.1117/1.NPh.3.3.031414. Epub 2016 Jul 12. PMID 27429995
- [Derived] Nguyen TTP, Hoang HB, Vu HTT. Effectiveness of multifaceted interventions including motivational interviewing and home-based rehabilitation program for improving mental and physical health in stroke patients: A randomized controlled trial. Int J Nurs Stud Adv. 2024 Oct 30;7:100259. doi: 10.1016/j.ijnsa.2024.100259. eCollection 2024 Dec. PMID 39610664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2021 to March 2022, individuals participating in the study were selected from the statistical list of stroke patients diagnosed by a neurologist at the National Geriatric Hospital.
Pre-assignment Details: Of 129 individuals assessed for eligibility (screened), 92 provided informed consent and were randomized (46 per arm). 37 were excluded due to not meeting the inclusion criteria, declining to participate, or other reasons.
Groups:
- Multi-intervention Program: A multi-intervention program will be designed for stroke patients, including:
  1. Periodic health check program for post-stroke: The stroke survivors will be assessed their physical and mental health, and harmful behaviors at 0, 1, 3, and 6 months by specific scales.
  2. Guiding the appropriate rehabilitation exercises: The appropriate rehabilitation exercises will be designed and guided for each patient and they will be followed up by the daily online report. This arm was performed in months 1+2 (once a week), months 3+4 (every 2 weeks), and months 5 + 6 (every 4 weeks).
  3. Motivational Interviewing will be conducted with post-stroke patients in the first month (once a week), the second month (every 2 weeks), and the third month (every 2 weeks). Each appointment will last for 1-2 hours. This intervention method aims to discover and resolve patients' conflicts through standardized communication skills to improve their mental health and change negative behaviors.
  4. Functional near-infrared spectroscopy: The fNIRS devices as an effective monitoring and therapeutic tool, evaluating the evolution of neural activity. Moreover, the cortex hemodynamic measure by fNIRS may detect early various mental disorders such as depression, fatigue, schizophrenia... through cognitive tasks.
- Standard Care: Standard health check and fNIRS measure
  1. Periodic health check program for post-stroke: The stroke survivors will be assessed their physical and mental health, and harmful behaviors at 0, 1, 3, and 6 months by specific scales.
  2. Functional near-infrared spectroscopy: The fNIRS devices as an effective monitoring and therapeutic tool, evaluating the evolution of neural activity. Moreover, the cortex hemodynamic measure by fNIRS may detect early various mental disorders such as depression, fatigue, schizophrenia... through cognitive tasks.
Period: Overall Study
Arm/Group | Multi-intervention Program | Standard Care
Started | 46 | 46
Completed | 37 | 43
Not Completed | 9 | 3
Not completed — At the time of confirming dropout, the dropout patients had not experienced any SAEs or fatalities. | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Multi-intervention Program: A multi-intervention program was designed for intervention groups, including:
  1. Periodic health check program for post-stroke: The stroke survivors will be assessed for their physical and mental health, and harmful behaviors at 0, 1, 3, and 6 months by specific scales.
  2. Guiding the appropriate rehabilitation exercises: The appropriate rehabilitation exercises will be designed and guided for each patient and they will be followed up by the daily online report. This arm was performed in months 1+2 (once a week), months 3+4 (every 2 weeks), and months 5 + 6 (every 4 weeks).
  3. Motivational Interviewing will be conducted with post-stroke patients in the first month (once a week), the second month (every 2 weeks), and the third month (every 2 weeks). Each appointment will last for 1-2 hours. This intervention method aims to discover and resolve patients' conflicts through standardized communication skills to improve their mental health and change negative behaviors.
  4. Functional near-infrared spectroscopy: The fNIRS devices as an effective monitoring and therapeutic tool, evaluating the evolution of neural activity. Moreover, the cortex hemodynamic measure by fNIRS may detect early various mental disorders such as depression, fatigue, and schizophrenia... through cognitive tasks.
- Standard Care: The control group received the standard health check and fNIRS measure:
  1. Periodic health check program for post-stroke: The stroke survivors will be assessed for their physical and mental health, and harmful behaviors at 0, 1, 3, and 6 months by specific scales.
  2. Functional near-infrared spectroscopy: The fNIRS devices as an effective monitoring and therapeutic tool, evaluating the evolution of neural activity. Moreover, the cortex hemodynamic measure by fNIRS may detect early various mental disorders such as depression, fatigue, schizophrenia... through cognitive tasks.
- Total: Total of all reporting groups
Arm/Group | Multi-intervention Program | Standard Care | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (10.2) | 69.8 (12.1) | 72.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 24 | 24 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Marital status [Count of Participants; unit: Participants]
  Living with spouse | 24 | 26 | 50
  Single, widow/widower | 22 | 20 | 42
Employment status [Count of Participants; unit: Participants]
  Inactive | 25 | 15 | 40
  Active | 21 | 31 | 52
Education [Count of Participants; unit: Participants]
  Secondary school & lower | 20 | 12 | 32
  High school & upper | 26 | 34 | 60
Body mass index (BMI) [Count of Participants; unit: Participants]
  Normal (18.5-24.9) | 28 | 29 | 57
  Overweight (25.0-29.9)/ Obese (≥30.0) | 18 | 17 | 35
Blood pressure [Count of Participants; unit: Participants]
  Normal (<140 mmHg/<90 mmHg) | 28 | 34 | 62
  High (≥140 mmHg and/or ≥90 mmHg) | 18 | 12 | 30
Poor sleep quality - Pittsburgh Sleep Quality Index [Count of Participants; unit: Participants]
  No | 8 | 16 | 24
  Yes | 38 | 30 | 68
Charlson Comorbidity Index (CCI) [Mean (Standard Deviation); unit: units on a scale] — Charlson Comorbidity Index (CCI) quantifies comorbidity burden using 17 conditions with weights 1, 2, 3, or 6. The total CCI score is the sum of weights of all present conditions (no double-counting of overlapping categories); possible range 0-33. Higher scores indicate greater comorbidity burden and worse prognosis. Baseline CCI was abstracted from medical records/ICD-10 by trained staff at enrollment. Unit: scores on a scale; values shown as mean (SD) by arm
  units on a scale | 5.7 (1.5) | 5.4 (1.4) | 5.6 (1.5)
Stroke classification [Count of Participants; unit: Participants]
  Ischemia | 21 | 15 | 36
  Hemorrhage | 5 | 7 | 12
  Unknown | 20 | 24 | 44
Frequency of stroke occurrences [Count of Participants; unit: Participants]
  Once | 34 | 31 | 65
  Twice or more | 12 | 15 | 27
Duration from stroke onset to participate in the study [Count of Participants; unit: Participants]
  1 month to < 3 months | 9 | 11 | 20
  3 months to < 6 months | 22 | 19 | 41
  6 months to 1 year | 15 | 16 | 31
Hemispheric lesion locations [Count of Participants; unit: Participants]
  Left-sided | 6 | 0 | 6
  Right-sided | 17 | 24 | 41
  Unknown | 23 | 22 | 45
Disability levels of stroke survivors - MRS [Count of Participants; unit: Participants]
  No symptoms (0) | 5 | 1 | 6
  No significant disability (1) | 9 | 12 | 21
  Slight disability (2) | 5 | 4 | 9
  Moderate disability (3) | 9 | 6 | 15
  Moderate-severe disability (4) | 18 | 23 | 41
National Institutes of Health Stroke Scale - NIHSS (score) [Mean (Standard Deviation); unit: units on a scale] — National Institutes of Health Stroke Scale (NIHSS) is a 15-item clinician-rated scale of neurological deficit (level of consciousness, gaze, visual fields, facial palsy, motor arm/leg, limb ataxia, sensory, language, dysarthria, extinction/inattention). Items are scored 0-2/3/4 as specified; the **total score is the sum of item scores, range 0-42. Higher scores indicate more severe neurological impairment (worse outcome); 0 = no deficit; 1-4 = minor; 5-15 = moderate; 16-20 = moderate-to-severe; 21-42 = severe.
  units on a scale | 5.9 (4.6) | 9.2 (6.4) | 7.6 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline Patient Health Questionnaire at 1, 3, and 6 Months
Description: The Patient Health Questionnaire-9 is a screening tool for post-stroke depression and assessing the changes at baseline, 1, 3, and 6 months. The possible range is 0-27 and the higher scores mean worse outcomes.
Time Frame: Baseline, 1, 3, and 6 months post intervention
Population: Over 6 months, the numbers of patients lost to follow-up in the intervention and control groups were respectively 9:0 (after 1 month), 9:0 (after 3 months), and 9:3 (after 6 months)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multi-intervention Program | Standard Care
Number analyzed (Participants) | 46 | 46
units on a scale
  Baseline | 10.9 (6.5) | 10.3 (5.9)
  After 1 month: number analyzed (Participants) | 37 | 46
  After 1 month | 9.1 (1.0) | 19.7 (3.8)
  After 3 months: number analyzed (Participants) | 37 | 46
  After 3 months | 3.1 (2.8) | 24.5 (2.8)
  After 6 months: number analyzed (Participants) | 37 | 43
  After 6 months | 1.8 (1.9) | 25.6 (2.9)
Statistical Analysis 1: Comparison: Multi-intervention Program vs Standard Care; We calculated that 92 participants randomized in a 1:1 fashion between the 2 groups would have at least 80% power to detect a difference of 3.43 points in mean score in improving physical and mental health after stroke (based on J.Sims et al in 2008) between intervention and control groups from baseline to the 6th month. The sample size was determined using a 2-sided 2-sample t-test (a=0.05). Assumptions included a common standard deviation of 5.49 and a discontinuation rate of 10%; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Median Difference (Net) = 0.6, 95% CI 2-sided [-1.9 to 3.2], Standard Error of Mean 1.3 — Treatment Difference = Intervention group - Control group; (1) Variables with multiple measurements over time were compared using the repeated measures ANOVA test to assess changes in Patient Health Questionnaire-9 score before and after intervention in two groups, calculating the time*group interaction; (2) Effect sizes after intervention are measured using Cohen's D, with values indicating small (d = 0.2), medium (d = 0.5), and large (d ≥ 0.8) effects

2. Primary Outcome: Fatigue Severity Scale (FSS)
Description: Fatigue Severity Scale (FSS) is a 9-item self-report questionnaire. Each item is rated 1 (strongly disagree) to 7 (strongly agree). The total score is the **sum of the 9 items (range 9-63); higher scores indicate greater fatigue severity (worse outcome). The total score (9-63) was analyzed at baseline, 1, 3, and 6 months. If ≤1 item was missing, the item was imputed per instrument guidance; otherwise the score was set to missing.
Time Frame: Baseline, 1, 3, and 6 months post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multi-intervention Program | Standard Care
Number analyzed (Participants) | 46 | 46
units on a scale
  Baseline | 35.2 (12.9) | 37.8 (11.4)
  After 1 month: number analyzed (Participants) | 37 | 46
  After 1 month | 28.5 (11.8) | 43.4 (8.7)
  After 3 months: number analyzed (Participants) | 37 | 46
  After 3 months | 17.8 (5.9) | 53.9 (8.1)
  After 6 months: number analyzed (Participants) | 37 | 43
  After 6 months | 14.4 (4.9) | 57.9 (7.6)
Statistical Analysis 1: Comparison: Multi-intervention Program vs Standard Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = -2.6, 95% CI 2-sided [-7.6 to 2.5], Standard Error of Mean 2.5 — Treatment Difference = Intervention group - Control group; (1) Variables with multiple measurements over time were compared using the repeated measures ANOVA test to assess changes in Fatigue Severity Scale score before and after intervention in two groups, calculating the time*group interaction; (2) Effect sizes after intervention are measured using Cohen's D, with values indicating small (d = 0.2), medium (d = 0.5), and large (d ≥ 0.8) effects

3. Primary Outcome: Changes From Baseline Mini-Mental State Examination at 1, 3, and 6 Months
Description: Mini-Mental State Examination is a screening tool for post-stroke cognitive impairment. Scores range from 0 to 30 points, with lower scores indicating greater impairment.
Time Frame: Baseline, 1, 3, and 6 month post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multi-intervention Program | Standard Care
Number analyzed (Participants) | 46 | 46
units on a scale
  Baseline | 16.2 (7.0) | 18.3 (8.9)
  After 1 month: number analyzed (Participants) | 37 | 46
  After 1 month | 13.5 (9.7) | 18.5 (8.7)
  After 3 months: number analyzed (Participants) | 37 | 46
  After 3 months | 17.9 (10.3) | 16.2 (7.6)
  After 6 months: number analyzed (Participants) | 37 | 43
  After 6 months | 19.5 (10.6) | 15.0 (8.3)
Statistical Analysis 1: Comparison: Multi-intervention Program vs Standard Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = -2.1, 95% CI 2-sided [-5.4 to 1.3], Standard Error of Mean 1.7 — Treatment Difference = Intervention group - Control group; (1) Variables with multiple measurements over time were compared using the repeated measures ANOVA test to assess changes in Mini-Mental State Examinationscore before and after intervention in two groups, calculating the time*group interaction; (2) Effect sizes after intervention are measured using Cohen's D, with values indicating small (d = 0.2), medium (d = 0.5), and large (d ≥ 0.8) effects

4. Primary Outcome: Changes From Baseline Barthel Index at 1, 3, and 6 Months
Description: Measure the changes of activities of daily living through assessing functional independence during half-year post-randomization. The score of the Barthel Index ranging from 0 to 100 was collected when 0 is the minimum (worst outcome) and 100 is the maximum (best outcome).
Time Frame: Baseline, 1, 3, and 6 months post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multi-intervention Program | Standard Care
Number analyzed (Participants) | 46 | 46
units on a scale
  Baseline | 55.5 (36.2) | 55.4 (34.3)
  After 1 month: number analyzed (Participants) | 37 | 46
  After 1 month | 58.8 (35.2) | 55.7 (33.9)
  After 3 months: number analyzed (Participants) | 37 | 46
  After 3 months | 68.8 (28.6) | 56.2 (33.3)
  After 6 months: number analyzed (Participants) | 37 | 43
  After 6 months | 68.8 (28.6) | 54.5 (33.0)
Statistical Analysis 1: Comparison: Multi-intervention Program vs Standard Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Over 6 months, the number of patients who losted to follow-up of intervention and control group were respectively 9:0 (after 1 month), 9:0 (after 3 months), and 9:3 (after 6 months); p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.1, 95% CI 2-sided [-14.5 to 14.7], Standard Error of Mean 7.4 — Treatment Difference = Intervention group - Control group; (1) Variables with multiple measurements over time were compared using the repeated measures ANOVA test to assess changes in Barthel Index score before and after intervention in two groups, calculating the time*group interaction; (2) Effect sizes after intervention are measured using Cohen's D, with values indicating small (d = 0.2), medium (d = 0.5), and large (d ≥ 0.8) effects

5. Primary Outcome: Changes From Baseline of Physical Domain - Stroke Impact Scale at 1, 3, and 6 Months
Description: The Stroke Impact Scale evaluates the post-stroke quality of life, utilizing a scoring system ranging from 0 to 100, higher scores denote improved quality of life. This scale consists of 08 domains, including (1) strength; (2) memory; (3) emotion; (4) communication; (5) activities of daily living independence; (6) mobility; (7) hand function; and (8) participation. The Physical domain was calculated from the domains by averaging the values (1+5+6+7)/4.
Time Frame: Baseline, 1, 3, and 6 months post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multi-intervention Program | Standard Care
Number analyzed (Participants) | 46 | 46
units on a scale
  Baseline | 36.9 (24.8) | 44.4 (29.3)
  After 1 month: number analyzed (Participants) | 37 | 46
  After 1 month | 28.4 (24.3) | 37.8 (28.0)
  After 3 months: number analyzed (Participants) | 37 | 46
  After 3 months | 34.7 (26.7) | 38.2 (27.7)
  After 6 months: number analyzed (Participants) | 37 | 43
  After 6 months | 38.5 (26.8) | 32.0 (27.3)
Statistical Analysis 1: Comparison: Multi-intervention Program vs Standard Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p < 0.05; Mean Difference (Net) = -7.6, 95% CI 2-sided [-18.8 to 3.7], Standard Error of Mean 5.6 — Treatment Difference = Intervention group - Control group; (1) Variables with multiple measurements over time were compared using the repeated measures ANOVA test to assess changes in Physical domain score of Stroke Impact Scale before and after intervention in two groups, calculating the time*group interaction; (2) Effect sizes after intervention are measured using Cohen's D, with values indicating small (d = 0.2), medium (d = 0.5), and large (d ≥ 0.8) effects

6. Secondary Outcome: Changes From Baseline of Stroke Impact Scale at 1, 3, and 6 Months
Description: The Stroke Impact Scale evaluates the post-stroke quality of life, utilizing a scoring system ranging from 0 to 100, higher scores denote improved quality of life. This scale consists of 08 domains, including (1) strength; (2) memory; (3) emotion; (4) communication; (5) activities of daily living independence; (6) mobility; (7) hand function; and (8) participation
Time Frame: Baseline, 1, 3, and 6 months post intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multi-intervention Program | Standard Care
Number analyzed (Participants) | 46 | 46
units on a scale
  Baseline | 45.4 (16.4) | 53.2 (19.2)
  After 1 month: number analyzed (Participants) | 37 | 46
  After 1 month | 48.3 (15.3) | 44.7 (19.6)
  After 3 months: number analyzed (Participants) | 37 | 46
  After 3 months | 58.5 (15.1) | 40.5 (19.2)
  After 6 months: number analyzed (Participants) | 37 | 43
  After 6 months | 62.6 (13.8) | 37.0 (18.8)
Statistical Analysis 1: Comparison: Multi-intervention Program vs Standard Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.05, t-test, 2 sided — The threshold for statistical significance was p = 0.05; Mean Difference (Net) = -7.8, 95% CI 2-sided [-15.2 to -0.3], Standard Error of Mean -3.7 — Treatment Difference = Intervention group - Control group; (1) Variables with multiple measurements over time were compared using the repeated measures ANOVA test to assess changes in Stroke Impact Scale score before and after intervention in two groups, calculating the time*group interaction; (2) Effect sizes after intervention are measured using Cohen's D, with values indicating small (d = 0.2), medium (d = 0.5), and large (d ≥ 0.8) effects

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Multi-intervention Program | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

LIMITATIONS AND CAVEATS:
Our study had several limitations as follows: Firstly, the small sample size limited a thorough exploration of underlying mechanisms. Secondly, participant heterogeneity may have influenced outcomes. Future research should employ more detailed recruitment methods. Lastly, the 6-month follow-up period may not fully capture the long-term impacts of the intervention. Further investigation is needed to assess sustainability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-12-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT04941482/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT04941482/SAP_001.pdf
  • Informed Consent Form (2021-12-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT04941482/ICF_002.pdf